CLINICAL TRIAL: NCT03524014
Title: Hepatitis E Infection : Emergence Mechanisms in North-Eastern France of Polymorphic Clinical Forms.
Acronym: VHENE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A00117-48
Record Dates: First submitted 2018-04-18; First posted 2018-05-14 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis E Infection in Humans and in Environment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HEV-infected patients with hepatitis
  Interventions: Other: Only advice for diagnosis and prevention
- HEV-infected patients with neurological features
  Interventions: Other: Only advice for diagnosis and prevention
- HEV-infected patients with kidney features
  Interventions: Other: Only advice for diagnosis and prevention

INTERVENTIONS:
Other: Only advice for diagnosis and prevention — Only advice for diagnosis and prevention

SUMMARY:
The present research aims to collect virological and clinical data on hepatitis E virus (HEV) infections, either in acute or chronic forms of HEV infection in North-Eastern France, with liver- or non liver-related symptoms, plus data on HEV circulation in the outside environment. The purpose of this study is to improve the diagnosis and care of HEV-infected patients, as well as the preventive features to take into account in order to avoid food- and environment-borne infections. At last, we will investigate HEV molecular characteristics, with the hypothesis that some advantageous HEV strains coul be more pathogenic for some tissues and/or organs.

ELIGIBILITY:
Inclusion Criteria:

* HEV-infected patients, with hepatitis and/or neurological and/or renal symptoms

Exclusion Criteria:

* Patients, with hepatitis and/or neurological and/or renal symptoms, infected by other viruses leading to hepatitis (hepatitis B, hepatitis C, hepatitis A ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusions during 2 years (2018-2019):
  * HEV infection, liver-related syndroms (either acute or chronic), n=20
  * HEV-infection, neurological (n=5; controls n=5) or renal syndroms (5-10; controls n= 5-10)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Anti-HEV IgM (qualitative assay); | 2 years
  Guidelines to improve HEV detection by using the 2 virological assays
HEV RNA (quantitative PCR assay) | 2 years
  Guidelines to improve HEV detection by using the 2 virological assays

CONTACTS AND LOCATIONS:
Locations (1):
- Schvoerer, Vandœuvre-lès-Nancy, France